CLINICAL TRIAL: NCT01935050
Title: A Guided Cognitive-Behavioral Self-Help Treatment for Depression in Parkinson's Disease
Brief Title: Guided Self-Help for Depression in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Roseanne D Dobkin, PhD, Associate Professor of Psychiatry, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013002798
Record Dates: First submitted 2013-05-29; First posted 2013-09-04 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Depression; Parkinson's Disease
Keywords: Depression; Parkinson's disease; Cognitive-Behavioral Treatment
MeSH Terms: conditions — Depression; Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Guided Cognitive-Behavioral Self-Help (Experimental): All participants will receive the experimental intervention: Guided Cognitive-Behavioral Self-Help. The 10 patient treatment modules will incorporate exercise, behavioral activation, thought monitoring and restructuring, relaxation training, worry control, and sleep hygiene. The four caregiver educational modules will provide caregivers with the skills needed to facilitate patients' practice of treatment techniques learned in session. For example, caregivers will be taught to help patients identify negative thoughts and replace them with more balanced alternatives and will be given tools to assist patients complete therapy goals (i.e., exercise, socializing).
  Interventions: Behavioral: Guided Cognitive-Behavioral Self-Help

INTERVENTIONS:
Behavioral: Guided Cognitive-Behavioral Self-Help — Participants will complete the study treatment at home. Bi-weekly telephone support will be provided by study staff.

SUMMARY:
The purpose of this project is to develop and pilot-test a guided cognitive-behavioral self-help program for mild-to-moderate depression in Parkinson's disease (dPD). We will pilot-test the guided self-help treatment on 20 people with PD and their caregivers. The manual will be revised based on participant feedback. Several feasibility measures regarding the guided self-help program (i.e., recruitment, retention, enjoyment, helpfulness, adherence) will also be assessed. Moreover, preliminary estimates of effect size for this guided self-help program will be calculated and used in future research. We hypothesize that people with PD will report decreases in depression, anxiety, and negative thoughts and improvements in quality life and sleep and that caregivers will report decreases in burden after participating in the guided self-help program

DETAILED DESCRIPTION:
To our knowledge, Cognitive-Behavioral self-help interventions remain unexplored for depression in PD to date. The results of this study will be used to support future treatment development efforts for depression and other psychiatric complications in PD that may improve the access to and quality of mental health care in this medical population.

ELIGIBILITY:
Inclusion Criteria:

1. Previous diagnosis of Parkinson's disease by a general neurologist or Movement Disorders Specialist
2. Clinically significant depression as determined by study staff
3. 35-85 years old
4. Stable medication regimen ≥ 6 weeks
5. No change in mental health treatment in past 2 months _

Exclusion Criteria:

1. Severe depressive symptoms
2. Suicidal plans or intent
3. Significant cognitive impairment
4. Significant motor fluctuations (i.e., ≥ 50% of the day)
5. Unstable medical conditions
6. Receiving CBT elsewhere

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The Hamilton Depression Rating Scale | 14 weeks
  A clinician-administered rating scale for depression

SECONDARY OUTCOMES:
Beck Depression Inventory | 14 weeks
  A self-report measure of depression
Hamilton Anxiety Rating Scale | 14 weeks
  A clinician-administered rating scale of anxiety
Inference Questionnaire | 14 weeks
  Self-report measure of negative thoughts
Caregiver Distress Scale | 14 weeks
  Self-report measure of caregiver stress
Insomnia Severity Index | 14 weeks
  Self-report sleep scale
Medical Outcomes Short Form | 14 weeks
  Self-report quality of life scale
Feasibility and adherence measures | 10 weeks
  Feasibility [Likert ratings (0-10) on the dimensions of readability, clarity, effort, enjoyment, fatigue, helpfulness, and progress regarding treatment materials] and adherence measures [a numerical rating regarding the % of recommended activities accomplished]
Clinical Global Impression-Improvement Scale | 14 weeks
  Clinician-rated scale of depression improvement

CONTACTS AND LOCATIONS:
Overall Officials: Roseanne D Dobkin, PhD, Principal Investigator — Rutgers Robert Wood Johnson Medical School
Locations (1):
- Rutgers University-Robert Wood Johnson Medical School, Piscataway, New Jersey, United States